CLINICAL TRIAL: NCT06584370
Title: Transatrial Pericardial Separation to Enhance the Safety of Subxiphoid Pericardial Access for Lariat Lariat Left Atrial Appendage Ligation
Brief Title: Transatrial Pericardial Separation to Enhance Safety of Subxiphoid Pericardial Access for Left Atrial Appendage Ligation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Adam Greenbaum, Co-Director, Structural Heart Disease Program, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8874
Record Dates: First submitted 2015-04-29; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Ligation; Pericardium; Epicardial Mapping; Heart Atria; Cardiac Surgical Procedures; Cardiac Catheterization; Pneumopericardium; Left Atrial Appendage Occlusion
MeSH Terms: conditions — Atrial Fibrillation; Pneumopericardium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pericardial insufflation with CO2 (Experimental): Intentional transatrial introduction of a microcatheter to insufflate the pericardium with carbon dioxide, to separate the walls of the pericardium
  Interventions: Procedure: Pericardial insufflation with carbon dioxide through a transatrial microcatheter

INTERVENTIONS:
Procedure: Pericardial insufflation with carbon dioxide through a transatrial microcatheter — Separate the walls of the pericardium by insufflating the pericardial space with carbon dioide.

SUMMARY:
We use a tiny catheter through the heart to separate the pericardium with gas. We expect this to improve the safety of the Lariat procedure.

DETAILED DESCRIPTION:
The Lariat suture device enables non-surgical exclusion of the left atrial appendage possibly to prevent thromboembolism and stroke in patients with atrial fibrillation. Subxiphoid needle access to the pericardium (a standard approach to enter the pericardial space surrounding the heart using a needle underneath the breastbone) during Lariat risks injury to the heart surface that requires surgical repair.

In this protocol the investigators propose test a new method to increase the safety of needle access to the pericardium. Before needle access, the investigators introduce a separate tiny catheter into the pericardium from inside the heart through a tiny hole. The investigators then inject gas to push the heart away from the pericardial needle. This reduces the risk of injuring the heart during the standard Lariat procedure.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing subxiphoid access to the "empty" pericardial space as part of a Lariat left atrial appendage exclusion procedure
* Age ≥ 21 years

Exclusion Criteria:

• Does not consent to participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Successful subxiphoid needle access without myocardial injury | Immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Cohn WE, Winkler JA, Tuzun E, Hjelle A, Bassett K, Ahmad A, Frazier OH. Contrast pericardiography facilitates intrapericardial navigation under fluoroscopy. Ann Thorac Surg. 2010 Nov;90(5):1537-40. doi: 10.1016/j.athoracsur.2010.06.025. PMID 20971258
- [Result] Rogers T, Ratnayaka K, Schenke WH, Faranesh AZ, Mazal JR, O'Neill WW, Greenbaum AB, Lederman RJ. Intentional right atrial exit for microcatheter infusion of pericardial carbon dioxide or iodinated contrast to facilitate sub-xiphoid access. Catheter Cardiovasc Interv. 2015 Aug;86(2):E111-8. doi: 10.1002/ccd.25698. Epub 2014 Oct 28. PMID 25315516